CLINICAL TRIAL: NCT03476460
Title: Efficacy of Oral Sodium Chloride vs iv Sodium Chloride in the Prevention of Contrast Nephropathy in Outpatients
Brief Title: Sodium Chloride and Contrast Nephropathy
Acronym: PNIC-Na
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Universitario Ramon y Cajal (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Ministerio de Sanidad, Servicios Sociales e Igualdad (Other Government)
Responsible Party: Principal Investigator, Luis Manzano Espinosa, MD, PhD, Chief of Internal Medicine department, Hospital Universitario Ramon y Cajal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EC11-132
Record Dates: First submitted 2018-03-17; First posted 2018-03-26 (Actual); Results first posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Kidney Failure, Chronic; Kidney Failure, Acute; Heart Failure; Diabetes
Keywords: Acute kidney failure; CT scan; Iodine contrast; Sodium chloride
MeSH Terms: conditions — Kidney Failure, Chronic; Acute Kidney Injury; Heart Failure; Diabetes Mellitus | interventions — Sodium Chloride

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral sodium chloride (Experimental): Patients will receive capsules of sodium chloride and free water ingestion (for each capsule of sodium chloride, patients will take 250 ml of water, assuring a minimum ingestion of 750 ml of water) in the 48 hours prior contrast injection. Patients will take capsules of sodium chloride at a dose of 100 mg/kg during 48 hours previous the injection of contrast (48, 40, 32, 24, 16, and 8 hours), at the moment of contrast injection and 12 hours after the injection of contrast.
  Interventions: Drug: Oral sodium chloride
- Intravenous sodium chloride (Active Comparator): Patients will receive at hospital 3 ml/Kg of sodium chloride 0.9%, one hour previous contrast injection and 2 ml/kg during the 4 hours after contrast injection.
  Interventions: Drug: Intravenous sodium chloride

INTERVENTIONS:
Drug: Oral sodium chloride — Patients will receive capsules of sodium chloride and free water ingestion (for each capsule of sodium chloride, with 250 ml of water, assuring a minimum ingestion of 750 ml of water) in the 48 hours prior contrast injection. Patients will take capsules of sodium chloride at a dose of 100 mg/kg during 48 hours previous the injection of contrast (48, 40, 32, 24, 16, and 8 hours), at the moment of contrast injection and 12 hours after the injection of contrast.
  Arms: Oral sodium chloride
Drug: Intravenous sodium chloride — Patients will receive at hospital 3 ml/Kg of sodium chloride 0.9%, one hour previous contrast injection and 2 ml/kg during the 4 hours after contrast injection.
  Arms: Intravenous sodium chloride

SUMMARY:
This phase II, open, non-inferiority, randomized and controlled clinical trial is aimed to ascertain the incidence of contrast nephropathy in outpatients undergoing CT scan with contrast.

Patients will be randomized to receive oral prophylaxis with capsules of sodium chloride and free water ingestion or prophylaxis with sodium chloride 0.9% intravenous solution.

The total dose (mmol) of sodium chloride will be the same regardless administration via. The contrast will be iodixanol.

Patients >65 years, of both sexes, with at least one of the following criteria: diabetes, stable heart failure or chronic kidney disease (estimated glomerular filtration rate between 30 and 60 ml/min), undergoing CT scan with contrast, and who give written informed consent, will be included in the study. Patients with estimated glomerular filtration rate <30 ml/min, serum potassium <3.5 mEq/L, infusion of iodine contrast in the previous 15 days, administration of nephrotoxic drugs in the previous 72 hours or expected in the following hours after contrast infusion, decompensated chronic conditions (heart failure, chronic obstructive pulmonary disease, hypertension), allergy to iodine contrast, or the presence of hyperchloremia or hypernatremia, will be excluded from the study.

Contrast nephropathy will be defined as the increase of serum creatinine >0.3 mg/dL from baseline, or the reduction of estimated glomerular filtration rate (MDRD-4) >25% from baseline, in the first 48 hours after contrast administration.

DETAILED DESCRIPTION:
This phase II, open, non-inferiority, randomized and controlled clinical trial is aimed to ascertain the incidence of contrast nephropathy in outpatients undergoing CT scan with contrast.

Patients will be randomized to receive oral prophylaxis with capsules of sodium chloride and free water ingestion or prophylaxis with sodium chloride 0.9% intravenous solution.

In those patients randomly allocated to oral prophylaxis (n=133), patients will receive capsules of sodium chloride and free water ingestion (for each capsule of sodium chloride, patients will take 250 ml of water, assuring a minimum ingestion of 750 ml of water) in the 48 hours prior contrast injection. Patients will take capsules of sodium chloride at a dose of 100 mg/kg during 48 hours previous the injection of contrast (48, 40, 32, 24, 16, and 8 hours), at the moment of contrast injection and 12 hours after the injection of contrast. In those patients randomly allocated to receive sodium chloride 0.9% intravenous solution (n=133), patients will receive at hospital 3 ml/Kg of sodium chloride 0.9%, one hour previous contrast injection and 2 ml/kg during the 4 hours after contrast injection. The total dose (mmol) of sodium chloride will be the same regardless administration via. The contrast will be iodixanol (320 mg of iodine/ml, in 100 ml, at an infusion rate of 2-5 ml/sec).

Patients >65 years, of both sexes, with at least one of the following criteria: diabetes, stable heart failure or chronic kidney disease (estimated glomerular filtration rate between 30 and 60 ml/min), undergoing CT scan with contrast, and who give written informed consent, will be included in the study. Patients with estimated glomerular filtration rate <30 ml/min, serum potassium <3.5 mEq/L, infusion of iodine contrast in the previous 15 days, administration of nephrotoxic drugs in the previous 72 hours or expected in the following hours after contrast infusion, decompensated chronic conditions (heart failure, chronic obstructive pulmonary disease, hypertension), allergy to iodine contrast, or the presence of hyperchloremia or hypernatremia, will be excluded from the study.

Contrast nephropathy will be defined as the increase of serum creatinine >0.3 mg/dL from baseline, or the reduction of estimated glomerular filtration rate (MDRD-4) >25% from baseline, in the first 48 hours after contrast administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients >65 years,
* Both sexes,
* With at least one of the following criteria: diabetes or stable heart failure or chronic kidney disease (estimated glomerular filtration rate between 30 and 60 ml/min),
* Undergoing CT scan with contrast
* Written informed consent.

Exclusion Criteria:

* Estimated glomerular filtration rate <30 ml/min,
* Serum potassium <3.5 mEq/L,
* Infusion of iodine contrast in the previous 15 days,
* Administration of nephrotoxic drugs in the previous 72 hours or expected in the following hours after contrast infusion,
* Decompensated chronic conditions (heart failure, chronic obstructive pulmonary disease, hypertension),
* Allergy to iodine contrast,
* Presence of hyperchloremia or hypernatremia.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 271 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2019-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luis Manzano, MD, PhD, Principal Investigator — Hospital Universitario Ramon y Cajal
Locations (1):
- Hospital Universitario Ramon y Cajal, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data Availability Statement The data presented in this study are available on request from the corresponding author. The data are not publicly available due to participant confidentiality.
Supporting Information: Study Protocol, ICF
Time Frame: After revision and approval of the principal investigator.
Access Criteria: Approval of the principal investigator.

REFERENCES:
- [Result] Suarez Carantona C, Escobar Cervantes C, Fabregate M, Lopez Rodriguez M, Bara Ledesma N, Soto Perez-Olivares J, Ruiz Ortega RA, Lopez Castellanos G, Olavarria Delgado A, Blazquez Sanchez J, Gomez Del Olmo V, Moralejo Martin M, Pumares Alvarez MB, Sanchez Gallego MC, Llacer P, Liano F, Manzano L. Oral Sodium Chloride in the Prevention of Contrast-Associated Acute Kidney Injury in Elderly Outpatients: The PNIC-Na Randomized Non-Inferiority Trial. J Clin Med. 2023 Apr 19;12(8):2965. doi: 10.3390/jcm12082965. PMID 37109303

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at Hospital Universitario Ramón y Cajal, Madrid, Spain, between April 2014 and November 2019.
Pre-assignment Details: A total of 271 patients were enrolled in the study, of whom 19 (7.0%) did not meet the criteria for per-protocol analysis and were therefore excluded from the main analysis. The reasons for exclusion included voluntary withdrawal (n=5), hospitalisation for bronchospasm (n=1), missing laboratory tests (n=10), and non-compliance with treatment (n=3). Thus, the main analysis (per-protocol) consisted of n=252 patients, of whom 123 received oral hydration and 129 received intravenous hydration.
Period: Overall Study
Arm/Group | Oral Sodium Chloride | Intravenous Sodium Chloride
Started | 134 | 137
Completed | 123 | 129
Not Completed | 11 | 8
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Non-compliance with treatment | 3 | 0
Not completed — Missing laboratory tests | 5 | 5
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Sodium Chloride | Intravenous Sodium Chloride | Total
Number analyzed (Participants) | 123 | 129 | 252
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.1 (6.1) | 74.6 (6.8) | 74.4 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 50 | 84
  Male | 89 | 79 | 168
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Spain | 123 | 129 | 252
Hypertension [Count of Participants; unit: Participants] | 94 | 98 | 192
Diabetes [Count of Participants; unit: Participants] | 87 | 97 | 184
Current smoker [Count of Participants; unit: Participants] | 5 | 9 | 14
Cancer [Count of Participants; unit: Participants] | 68 | 59 | 127
Chronic kidney disease [Count of Participants; unit: Participants] | 53 | 47 | 100
Heart failure [Count of Participants; unit: Participants] | 16 | 25 | 41
Peripheral artery disease [Count of Participants; unit: Participants] | 11 | 8 | 19
Estimated glomerular filtration rate (eGFR) according to MDRD-4 [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 66.6 (19.4) | 69.0 (19.6) | 67.8 (19.5)
Serum creatinine [Mean (Standard Deviation); unit: mg/dL] | 1.09 (0.31) | 1.02 (0.29) | 1.06 (0.30)
Cystatin C [Mean (Standard Deviation); unit: mg/dL] | 1.36 (0.39) | 1.41 (0.46) | 1.38 (0.43)
Albumin-to-creatinine ratio [Median (Inter-Quartile Range); unit: mg/g] | 17.4 [10.1 to 81.9] | 19.4 [8.3 to 61.0] | 19.0 [8.8 to 66.3]
Urea [Mean (Standard Deviation); unit: mg/dL] | 49.1 (16.2) | 46.7 (18.8) | 47.8 (17.6)
Serum sodium [Mean (Standard Deviation); unit: mg/dL] | 139.2 (2.6) | 139.6 (3.1) | 139.4 (2.9)
Serum potassium [Mean (Standard Deviation); unit: mg/dL] | 4.5 (0.4) | 4.5 (0.5) | 4.5 (0.5)
B-type natriuretic peptide (BNP) [Median (Inter-Quartile Range); unit: pg/mg] | 56.6 [24.4 to 153.5] | 54.0 [29.6 to 100.3] | 55.9 [27.9 to 119.9]
Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 13.6 (1.8) | 13.7 (1.7) | 13.6 (1.8)
Non-diuretic antihypertensives [Count of Participants; unit: Participants] | 95 | 97 | 192
Non-insulin antidiabetic drugs [Count of Participants; unit: Participants] | 81 | 86 | 167
Lipid-lowering agents [Count of Participants; unit: Participants] | 76 | 79 | 155
Diuretics [Count of Participants; unit: Participants] | 48 | 45 | 93
Body mass index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] | 23.0 (3.9) | 23.0 (3.7) | 23.0 (3.8)
Systolic blood pressure (SBP) [Mean (Standard Deviation); unit: mmHg] | 140.2 (19.8) | 143.1 (20.2) | 141.7 (20.0)
Heart rate [Mean (Standard Deviation); unit: bpm] | 71.1 (13.9) | 70.9 (11.1) | 71.0 (12.6)
Peripheral oxygen saturation (spO2) [Mean (Standard Deviation); unit: percentage of hemoglobin saturation] | 95.8 (2.4) | 95.4 (3.0) | 95.6 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acute Kidney Injury During the First 48 Hours After Contrast Administration
Description: Contrast-Associated Acute Kidney Injury, defined as the increase of serum creatinine >0.3 mg/dL from baseline, or the reduction of estimated glomerular filtration rate (MDRD-4) >25%, within 48h after contrast administration
Time Frame: Within 48h after contrast administration
Population: Per-protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Sodium Chloride | Intravenous Sodium Chloride
Number analyzed (Participants) | 123 | 129
Participants | 5 | 4
Statistical Analysis 1: Comparison: Oral Sodium Chloride vs Intravenous Sodium Chloride; Sample size was calculated to assess the non-inferiority of oral compared to intravenous hydration. We expected a primary outcome rate of 7% in the intravenous arm. We considered a priori a difference of no more than 5% in the incidence of CA-AKI in the oral compared to the intravenous arm (non-inferiority margin) to be acceptable. Thus, 266 participants, 133 per arm, were required to ensure at least 80% power at a significance level of α = 2.5% (one-sided); Test type: Non-Inferiority — We considered a priori a difference of no more than 5% in the incidence of CA-AKI in the oral compared to the intravenous arm (non-inferiority margin) to be acceptable. The non-inferiority of oral hydration would be shown if the upper limit of the 95% CI of the absolute risk difference between the groups was less than 5% (non-inferiority margin, indicated by the black dashed line); Risk Difference (RD) = 1.0, 95% CI 2-sided [-4.8 to 7.0] — The 95% confidence interval for the difference between the two independent proportions was calculated according to Wilson's method

2. Secondary Outcome: Estimated Glomerular Filtration Rate (eGFR) at 24h From Baseline
Description: Estimated glomerular filtration rate (eGFR) according to MDRD-4 at 24 hours from contrast administration (baseline), as an secondary efficacy laboratory assessment.
Time Frame: 24 hours from contrast administration (baseline)
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Oral Sodium Chloride | Intravenous Sodium Chloride
Number analyzed (Participants) | 123 | 129
mL/min/1.73 m^2 | 66.4 (18.9) | 68.8 (18.9)
Statistical Analysis 1: Comparison: Oral Sodium Chloride vs Intravenous Sodium Chloride; Comparison between means of both arms at 24h from baseline; Test type: Superiority; p = 0.299, t-test, 2 sided — A p-value <0.05 (two-sided) was considered for statistical significance

3. Secondary Outcome: Estimated Glomerular Filtration Rate (eGFR) at 48h From Baseline
Description: Estimated glomerular filtration rate (eGFR) according to MDRD-4 at 48 hours from contrast administration (baseline), as an secondary efficacy laboratory assessment.
Time Frame: 48 hours from contrast administration (baseline)
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Oral Sodium Chloride | Intravenous Sodium Chloride
Number analyzed (Participants) | 123 | 129
mL/min/1.73 m^2 | 66.1 (19.7) | 67.9 (19.6)
Statistical Analysis 1: Comparison: Oral Sodium Chloride vs Intravenous Sodium Chloride; Comparison between means of both arms at 48h from baseline; Test type: Superiority; p = 0.477, t-test, 2 sided — A p-value <0.05 (two-sided) was considered for statistical significance

4. Secondary Outcome: Serum Creatinine at 24h From Baseline
Description: Serum creatinine at 24 hours from contrast administration (baseline), as an secondary efficacy laboratory assessment.
Time Frame: 24 hours from contrast administration (baseline)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Oral Sodium Chloride | Intravenous Sodium Chloride
Number analyzed (Participants) | 123 | 129
mg/dL | 1.10 (0.33) | 1.02 (0.29)
Statistical Analysis 1: Comparison: Oral Sodium Chloride vs Intravenous Sodium Chloride; Test type: Superiority — Comparison between means of both arms at 24h from baseline; p = 0.042, t-test, 2 sided — A p-value <0.05 (two-sided) was considered for statistical significance

5. Secondary Outcome: Serum Creatinine at 48h From Baseline
Description: Serum creatinine at 48 hours from contrast administration (baseline), as an secondary efficacy laboratory assessment.
Time Frame: 48 hours from contrast administration (baseline)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Oral Sodium Chloride | Intravenous Sodium Chloride
Number analyzed (Participants) | 123 | 129
mg/dL | 1.10 (0.36) | 1.04 (0.31)
Statistical Analysis 1: Comparison: Oral Sodium Chloride vs Intravenous Sodium Chloride; Test type: Superiority — Comparison between means of both arms at 48h from baseline; p = 0.121, t-test, 2 sided — A p-value <0.05 (two-sided) was considered for statistical significance

6. Secondary Outcome: Cystatin C at 24h From Baseline
Description: Cystatin C at 24 hours from contrast administration (baseline), as an secondary efficacy laboratory assessment.
Time Frame: 24 hours from contrast administration (baseline)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Oral Sodium Chloride | Intravenous Sodium Chloride
Number analyzed (Participants) | 123 | 129
mg/dL | 1.38 (0.44) | 1.33 (0.46)
Statistical Analysis 1: Comparison: Oral Sodium Chloride vs Intravenous Sodium Chloride; Test type: Superiority — Comparison between means of both arms at 24h from baseline; p = 0.418, t-test, 2 sided — A p-value <0.05 (two-sided) was considered for statistical significance

7. Secondary Outcome: Cystatin C at 48h From Baseline
Description: Cystatin C at 48 hours from contrast administration (baseline), as an secondary efficacy laboratory assessment.
Time Frame: 48 hours from contrast administration (baseline)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Oral Sodium Chloride | Intravenous Sodium Chloride
Number analyzed (Participants) | 123 | 129
mg/dL | 1.36 (0.43) | 1.36 (0.46)
Statistical Analysis 1: Comparison: Oral Sodium Chloride vs Intravenous Sodium Chloride; Test type: Superiority — Comparison between means of both arms at 24h from baseline; p = 0.901, t-test, 2 sided — A p-value <0.05 (two-sided) was considered for statistical significance

8. Secondary Outcome: Albumin-to-creatinine Ratio at 24h From Baseline
Description: Albumin-to-creatinine ratio at 24 hours from contrast administration (baseline), as an secondary efficacy laboratory assessment.
Time Frame: 24 hours from contrast administration (baseline)
Measure: Median (Inter-Quartile Range); unit: mg/g
Arm/Group | Oral Sodium Chloride | Intravenous Sodium Chloride
Number analyzed (Participants) | 123 | 129
mg/g | 17.2 [8.3 to 72.0] | 17.0 [9.3 to 65.5]
Statistical Analysis 1: Comparison: Oral Sodium Chloride vs Intravenous Sodium Chloride; Test type: Superiority — Comparison between means of both arms at 24h from baseline; p = 0.720, Wilcoxon (Mann-Whitney) — A p-value <0.05 (two-sided) was considered for statistical significance

9. Secondary Outcome: Albumin-to-creatinine Ratio at 48h From Baseline
Description: Albumin-to-creatinine ratio at 48 hours from contrast administration (baseline), as an secondary efficacy laboratory assessment.
Time Frame: 48 hours from contrast administration (baseline)
Measure: Median (Inter-Quartile Range); unit: mg/g
Arm/Group | Oral Sodium Chloride | Intravenous Sodium Chloride
Number analyzed (Participants) | 123 | 129
mg/g | 17.6 [9.0 to 69.2] | 18.2 [9.0 to 50.1]
Statistical Analysis 1: Comparison: Oral Sodium Chloride vs Intravenous Sodium Chloride; Test type: Superiority — Comparison between means of both arms at 48h from baseline; p = 0.688, Wilcoxon (Mann-Whitney) — A p-value <0.05 (two-sided) was considered for statistical significance

10. Secondary Outcome: Urea at 24h From Baseline
Description: Urea at 24 hours from contrast administration (baseline), as an secondary efficacy laboratory assessment.
Time Frame: 24 hours from contrast administration (baseline)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Oral Sodium Chloride | Intravenous Sodium Chloride
Number analyzed (Participants) | 123 | 129
mg/dL | 43.7 (18.7) | 42.2 (18.2)
Statistical Analysis 1: Comparison: Oral Sodium Chloride vs Intravenous Sodium Chloride; Test type: Superiority — Comparison between means of both arms at 24h from baseline; p = 0.535, t-test, 2 sided — A p-value <0.05 (two-sided) was considered for statistical significance

11. Secondary Outcome: Urea at 48h From Baseline
Description: Urea at 48 hours from contrast administration (baseline), as an secondary efficacy laboratory assessment.
Time Frame: 48 hours from contrast administration (baseline)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Oral Sodium Chloride | Intravenous Sodium Chloride
Number analyzed (Participants) | 123 | 129
mg/dL | 46.0 (19.5) | 43.5 (20.1)
Statistical Analysis 1: Comparison: Oral Sodium Chloride vs Intravenous Sodium Chloride; Test type: Superiority — Comparison between means of both arms at 48h from baseline; p = 0.338, t-test, 2 sided — A p-value <0.05 (two-sided) was considered for statistical significance

12. Secondary Outcome: Serum Sodium at 24h From Baseline
Description: Serum sodium at 24 hours from contrast administration (baseline), as an secondary efficacy laboratory assessment.
Time Frame: 24 hours from contrast administration (baseline)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Oral Sodium Chloride | Intravenous Sodium Chloride
Number analyzed (Participants) | 123 | 129
mg/dL | 139.4 (2.6) | 139.3 (2.6)
Statistical Analysis 1: Comparison: Oral Sodium Chloride vs Intravenous Sodium Chloride; Test type: Superiority — Comparison between means of both arms at 24h from baseline; p = 0.764, t-test, 2 sided — A p-value <0.05 (two-sided) was considered for statistical significance

13. Secondary Outcome: Serum Sodium at 48h From Baseline
Description: Serum sodium at 48 hours from contrast administration (baseline), as an secondary efficacy laboratory assessment.
Time Frame: 48 hours from contrast administration (baseline)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Oral Sodium Chloride | Intravenous Sodium Chloride
Number analyzed (Participants) | 123 | 129
mg/dL | 139.2 (2.7) | 139.4 (2.6)
Statistical Analysis 1: Comparison: Oral Sodium Chloride vs Intravenous Sodium Chloride; Test type: Superiority — Comparison between means of both arms at 48h from baseline; p = 0.458, t-test, 2 sided — A p-value <0.05 (two-sided) was considered for statistical significance

14. Secondary Outcome: Serum Potassium at 24h From Baseline
Description: Serum potassium at 24 hours from contrast administration (baseline), as an secondary efficacy laboratory assessment.
Time Frame: 24 hours from contrast administration (baseline)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Oral Sodium Chloride | Intravenous Sodium Chloride
Number analyzed (Participants) | 123 | 129
mg/dL | 4.4 (0.4) | 4.4 (0.5)
Statistical Analysis 1: Comparison: Oral Sodium Chloride vs Intravenous Sodium Chloride; Test type: Superiority — Comparison between means of both arms at 24h from baseline; p = 0.893, t-test, 2 sided — A p-value <0.05 (two-sided) was considered for statistical significance

15. Secondary Outcome: Serum Potassium at 48h From Baseline
Description: Serum potassium at 48 hours from contrast administration (baseline), as an secondary efficacy laboratory assessment.
Time Frame: 48 hours from contrast administration (baseline)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Oral Sodium Chloride | Intravenous Sodium Chloride
Number analyzed (Participants) | 123 | 129
mg/dL | 4.4 (0.4) | 4.5 (0.5)
Statistical Analysis 1: Comparison: Oral Sodium Chloride vs Intravenous Sodium Chloride; Test type: Superiority — Comparison between means of both arms at 48h from baseline; p = 0.645, t-test, 2 sided — A p-value <0.05 (two-sided) was considered for statistical significance

ADVERSE EVENTS:
Time Frame: Within 48 hours from contrast administration (baseline).
Description: Adverse events were registered, including severity and relationship with study medication.
Arm/Group | Oral Sodium Chloride | Intravenous Sodium Chloride
All-Cause Mortality (participants affected / at risk) | 0/134 | 0/137
Serious Adverse Events (participants affected / at risk) | 0/134 | 0/137
Other Adverse Events (participants affected / at risk) | 31/134 | 6/137
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Sodium Chloride (N=134) | Intravenous Sodium Chloride (N=137)
Nausea (Gastrointestinal disorders) | 13 | 0
Vomiting (Gastrointestinal disorders) | 10 | 0
Abdominal discomfort (Gastrointestinal disorders) | 3 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Malaise/asthenia (General disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 0
Leg cramps (Musculoskeletal and connective tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Allergic reaction to contrast (Immune system disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chest tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Infection (Infections and infestations) | 0 | 1

LIMITATIONS AND CAVEATS:
The incidence of CA-AKI was much lower than expected at the time of study design. The definition of CA-AKI considered in our study is slightly different from that proposed in the clinical guidelines for AKI. Serial measurements of serum and urinary osmolality were not available in our trial. The trial was a single-center study, which might limit its external validity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-08-02): https://cdn.clinicaltrials.gov/large-docs/60/NCT03476460/Prot_SAP_000.pdf